CLINICAL TRIAL: NCT00191516
Title: An Open-Label Study on Effectiveness and Tolerability of Atomoxetine as Perceived by Patients, Parents, and Physicians in Children With Attention-Deficit/Hyperactivity Disorder in Germany
Brief Title: An Open-Label Study of Atomoxetine in Children With Attention-Deficit/Hyperactivity Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9496; B4Z-SB-LYDD
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: Atomoxetine

SUMMARY:
A single arm, open-label, phase 3 multicenter study to evaluate the effectiveness and tolerability of atomoxetine (given once daily, target dose 1.2 mg/kg/day), as perceived by patients, parents and physicians, and its impact on quality of sleep in children (aged 6 through 11 years) with Attention-Deficit/Hyperactivity Disorder treated as outpatients in Germany. An 8-week treatment phase is followed by a 16-week extension period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients who are at least 6 years of age and who will not have reached their 12th birthday
* Diagnosis of ADHD
* Normal intelligence

Exclusion Criteria:

* Weigh less than 20 kg or more than 60 kg at study entry
* Other relevant psychiatric diagnoses
* Are at serious suicidal risk as determined by the investigator
* Have a history of severe allergies
* Alcohol or drug abuse within the past 3 months

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 257
Dates: Start 2004-10; Study Completion 2006-02

PRIMARY OUTCOMES:
Global Impression of Perceived Difficulties (GIPD) scale at baseline, Week 8 and Week 24

SECONDARY OUTCOMES:
Pediatric Adverse Events Rating Scale (PAERS) during 8 and 24 weeks of treatment.
O'Brien Sleep Questionnaire during 8 and 24 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Chair — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cologne, Germany

REFERENCES:
- [Derived] Wehmeier PM, Schacht A, Dittmann RW, Banaschewski T. Minor differences in ADHD-related difficulties between boys and girls treated with atomoxetine for attention-deficit/hyperactivity disorder. Atten Defic Hyperact Disord. 2010 Jun;2(2):73-85. doi: 10.1007/s12402-010-0022-2. Epub 2010 Mar 30. PMID 21432592